CLINICAL TRIAL: NCT02461251
Title: Thromboelastometry-guided Treatment Protocol Versus Standard Care of Major Haemorrhage in Obstetric Patients
Acronym: ROTEM-PPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETL R15054
Record Dates: First submitted 2015-05-29; First posted 2015-06-03 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Obstetric Labor Complications; Hemorrhage
Keywords: Thromboelastometry; Obstetric Hemorrhage; Blood Component Transfusion
MeSH Terms: conditions — Obstetric Labor Complications; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotational thromboelastometry (ROTEM) (Experimental): Rotational thromboelastometry results are used to guide the treatment of major obstetric hemorrhage, eg. administration of prothrombin complex concentrate, fresh-frozen plasma, fibrinogen concentrate or platelets. In case of massive hemorrhage, "shock packs" of blood products in 1:1:1 ratio are administered.
  Interventions: Device: Rotational Thromboelastometry (ROTEM)
- Standard care (No Intervention): Patients are treated according to clinical decision making and conventional coagulation tests, and in case of massive hemorrhage, "shock packs" are administered.

INTERVENTIONS:
Device: Rotational Thromboelastometry (ROTEM) — A Point-of-care blood coagulation test tool is used to guide the treatment of major obstetric bleeding.
  Arms: Rotational thromboelastometry (ROTEM)

SUMMARY:
This is a prospective, randomized and controlled study to find out if a rotational thromboelastometry(ROTEM) guided treatment protocol reduces the need for blood transfusions in major obstetric haemorrhage compared to standard care of clinical decision making, conventional coagulation tests and massive transfusion protocol. Secondary aim is to find out if ROTEM can predict the incidence of thromboembolic events in this patient group.

DETAILED DESCRIPTION:
A comparison of two different treatment protocols is made in patients suffering major obstetric haemorrhage: those who after a normal delivery are bleeding more than 1000 ml and are in need of surgical intervention to control the bleeding and those in cesarean section with ongoing bleeding of more than 1000 ml. Patients are randomized in to two groups: the control group(n=30) will be treated according to a protocol based on clinical decision making, standard coagulation tests and massive transfusion packages of blood products(1:1:1), if needed. This is referred as 'Standard care' in this hospital. The intervention group(n=30) will be treated according to a rotational thromboelastometry guided protocol, and massive transfusion packages, if needed. The study is powered to detect a reduction of one unit in red blood cell transfusion. Blood product, fibrinogen concentrate, prothrombin complex concentrate usage and total amount of blood loss will be compared, and the number of transfusion related side effects and thromboembolic events 30 days after the bleeding will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Severe post-partum haemorrhage ie. active bleeding of more than 1000ml within 24 hours after vaginal delivery or cesarean section
* Informed consent (after randomization)

Exclusion Criteria:

* Known hemophilia or von Willebrand's disease
* Unacceptance of allogeneic blood products(Jehovah's witnesses)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2016-01; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Reduction in blood transfusions | 24 h

SECONDARY OUTCOMES:
Reduction of transfusion related side-effects | 30 days
Number of thromboembolic events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kuitunen, MD, PhD, Study Director — Tampere University Hospital; Samuli Jokinen, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jokinen S, Kuitunen A, Uotila J, Yli-Hankala A. Thromboelastometry-guided treatment algorithm in postpartum haemorrhage: a randomised, controlled pilot trial. Br J Anaesth. 2023 Feb;130(2):165-174. doi: 10.1016/j.bja.2022.10.031. Epub 2022 Dec 7. PMID 36496259